CLINICAL TRIAL: NCT05662176
Title: The Effect of Supportive Care Based on Trauma Informed Care at Childbirth on Perinatal Mental Health Outcomes: a Randomized Controlled Study
Brief Title: The Effect of Trauma Informed Care in Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gozde Gokce Isbir, Associate Prof, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DND
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Psychological Well-being; Childbirth; Care Pattern, Maternal
Keywords: Intrapartum supportive care; Trauma Informed Care; birth trauma; fear of childbirth; perinatal well-being
MeSH Terms: conditions — Psychological Well-Being; Birth Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Supportive Care based on trauma informed care (Experimental): Participants were provided care in different rooms, blinded to the differences in practice used between the two groups. In the same clinic, a room was designed as a positive delivery room by the researchers and a relaxing environment was created. In this room, supportive care based on trauma informed care was provided to the experimental group during birth.
  Interventions: Other: Experimental: Supportive Care based on trauma informed care
- Control: Standart care (Other): Participants in the control group, on the other hand, received the routine care given in the hospital by other midwives in the clinic, and there was a change of caregiver midwife during shift changes. The care provided in the hospital during delivery is mostly focused on low level of physical comfort and high level of follow-up.
  Interventions: Other: Standart care

INTERVENTIONS:
Other: Experimental: Supportive Care based on trauma informed care — Participants were provided care in different rooms, blinded to the differences in practice used between the two groups. In the same clinic, a room was designed as a positive delivery room by the researchers and a relaxing environment was created. In this room, supportive care based on trauma informed care was provided to the experimental group during birth.
  Arms: Experimental: Supportive Care based on trauma informed care
Other: Standart care — Participants in the control group, on the other hand, received the routine care given in the hospital by other midwives in the clinic, and there was a change of caregiver midwife during shift changes. The care provided in the hospital during delivery is mostly focused on low level of physical comfort and high level of follow-up.
  Arms: Control: Standart care

SUMMARY:
The aim of this study is to determine the effect of supportive care based on trauma informed care during childbirth on perinatal mental health outcomes.

DETAILED DESCRIPTION:
This is a randomized control experimental study. Data were collected from 100 women who attended supportive care based on trauma informed care or standart care from Turkey between July 2022 and September 2022. Participants who met the inclusion criteria were informed about the purpose of the study and the procedures to be performed, informed consent was obtained from those who agreed to participate, and women were assigned to the groups in line with a computer-based randomization program with an allocation ratio of 1:1. Block randomization could not be performed because of the different and long delivery processes. Data were collected in both groups at birth (latent phase, active phase, and transitional phase), within 24 hours of birth, and 6th-8th postpartum days after hospital admission and at least one hour of care. collected by the first author. The CONSORT directive was followed in the planning, implementation and writing of the research.

ELIGIBILITY:
Inclusion Criteria:

* The ages of 18-40 women,
* At least primary school graduate,
* Mother tongue Turkish,
* Single fetus,
* Term,
* Spontaneous birth,
* Cervical dilatation between 0-5 cm (latent phase) and without a condition that could prevent vaginal delivery.
* Primiparous women
* Not have any disease or complication and agreed to participate in the study were included.

Exclusion Criteria:

* Women who developed a complication with the fetus or themselves during delivery,
* Not be reached during follow-ups by telephone,
* Wanted to withdraw from the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2022-07-31 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Labor pain | through delivery, an average of 24th hours
  Women's labor pain at the time of birth were evaluated with the Visual Analogue Scale (DFS). The individual evaluates pain between "0-10 points. 0- I don't have any pain", "10- I have so much pain that I can't stand it". The higher the pain, the higher the score.
Fear of Childbirth (DFS) | through delivery, an average of 24th hours
  Women's fears at the time of birth were evaluated with the Delivery fear scale (DFS).
  This scale was developed for fear during delivery. The Turkish validity and reliability of the scale were performed. This scale consisting of 10 items is a 10-point Likert-type. The positive-meaning items are scored in reverse order. Therefore, the scores ranged from 10 to 100. The scale has no cutoff score, and high scores indicated higher fear.
Perceived control and support in birth (SCIB) | Postpartum 24th hours
  Women's perceptions of support and control at the time of birth were evaluated with the Perceived control and support in birth scale.
  SCIB was developed to measure perceived support and control in birth. The Turkish validity and reliability of the scale were performed. This scale consisting of 33 items is a 5-pointLikert-type (5 = agree completely to 1 = disagree completely). Ten items are scored in reverse order. The scores ranged from 33 to 165. SCIB subscales include internal control, external control, and support. The scale has no cutoff score, higher scores are associated with a higher degree of perceived support and of control during birth. The Cronbach's alpha for the original scale was measured as .95 and Turkish version was measured as 0.84. In this study, this scale was administered within 24 hours postpartum.
Birth Trauma (City BITS) | Postpartum 8 th week
  Birth trauma of women were evaluated with the City Birth Trauma Scale. City BiTS was developed to measure birth trauma. The Turkish validity and reliability of the scale were performed. The scale is a fourpoint Likert-type instrument composed of 29 items. Higher scores reflect greater risk for Post-traumatic Stress Disorder (PTSD). The Cronbach's alpha for the original scale was measured as .92 and Turkish version was measured as 0.91. In this study, 6-8 days after birth to determine whether they meet the criteria for birth trauma and birth-related PTSD.

CONTACTS AND LOCATIONS:
Locations (1):
- Gozde Gokce Isbir, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No